CLINICAL TRIAL: NCT04709445
Title: Objective Perfusion Rate Assessment of Gastrointestinal Anastomoses by Inflow and Outflow Analysis of Near-infrared Fluorescence Agents
Brief Title: Perfusion Rate Assessment by Near-infrared Fluorescence in Gastrointestinal Anastomoses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Benjamin Weixler, Attending Physician, Assistant Professor, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EA1/087/20
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Bowel Obstruction; Bowel Ischemia; Diverticulitis; Abnormality of the Gastrointestinal Tract; Symptomatic Disorders of the Gastrointestinal Tract; Stoma Ileostomy; Cancer of the Gastrointestinal Tract; Crohn Disease; Ulcerative Colitis; Familial Adenomatous Polyposis; Pancreatic Neoplasms; Hepatobiliary Neoplasm
Keywords: indocyanine green; objective perfusion rate; near infrared fluorescence; anastomotic leak; image guided surgery; anastomosis; perfusion assessment
MeSH Terms: conditions — Intestinal Obstruction; Diverticulitis; Gastrointestinal Neoplasms; Crohn Disease; Colitis, Ulcerative; Adenomatous Polyposis Coli; Pancreatic Neoplasms; Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: This is a non-randomised prospective cohort study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG-NIRF Imaging and objective perfusion rate (Experimental): Intraoperatively, ICG-NIRF imaging is used to visualize the blood supply and the rate of tissue perfusion in the area of the anastomotic site. Postoperatively, an additional ingress and egress analysis at specific regions of interest is performed.
  Interventions: Diagnostic Test: ICG-NIRF Imaging plus ingress and egress analysis

INTERVENTIONS:
Diagnostic Test: ICG-NIRF Imaging plus ingress and egress analysis — intraoperative NIRF Imaging using the fluorescence agent ICG (indocyanine-green) before and after anastomosis formation, postoperative analysis of ingress and egress for specific regions of interest

SUMMARY:
In this prospective, non-randomized cohort study, real-time intraoperative visualization using near-infrared-fluorescence by indocyanine green injection (ICG-NIRF) is performed at two to three time points during procedures of upper GI, lower GI and hepatobiliary surgery with anastomosis formation in open or laparoscopic surgery. Postoperatively, a detailed software-based assessment of each recording is performed to determine the objective ICG-NIRF perfusion rate before and after anastomosis formation, which is then correlated with the 30 day postoperative clinical outcome including occurrence of anastomotic leak.

DETAILED DESCRIPTION:
Near-infrared-fluorescence by indocyanine green (ICG-NIRF) utilises the fluorescent property of intravenously injected indocyanine green (ICG) as an intravascular indicator of tissue and bowel perfusion.

The investigators hypothesise that ICG-NIRF is a suitable, reliable and precise method of visualisation of the blood supply and bowel perfusion in the area of gastrointestinal and hepatobiliary anastomosis formation.

In this prospective, non-randomized cohort study, the respective upper GI, lower GI or hepatobiliary procedure with anastomosis is performed according to standard of care and indication for the corresponding disease including non-malignant, malignant and inflammatory conditions. The following procedures are included in the study, in open or laparoscopic surgery, according to the surgeon's choice:

Upper GI surgery:

* Esophageal resection
* Subtotal or total gastrectomy with or without jejunal pouch reconstruction
* Y-Roux-reconstruction
* Right or left colonic interposition (iso- or antiperistaltic)

Lower GI surgery:

* Jejunal or ileal segmental resection
* Ileal / Ileocoecal resection
* Colectomy with restorative ileal pouch formation and ileal-pouch-anal anastomosis
* Left or right-sided hemicolectomy
* Sigmoid resection
* Rectal resections (lower anterior resection (LAR), proctectomy with colo-anal anastomosis, abdominoperineal resection)
* Stoma closure

Hepatobiliary surgery:

- Pancreaticoduodenectomy

Written informed consent for participation and ICG-administration is obtained one day before surgery.

Intraoperatively, Indocyanine Green (ICG, VerDye, Diagnostic Green GmbH, Aschheim Germany, 25 mg vials) is dissolved in 5 mL sterile water to yield a 5 mg/mL concentration. It will then be administered intravenously at three consecutive time points as a bolus of 2 ml per time point at the most. The overall dose of ICG will amount to no more than 30mg of ICG per patient.

Real-time intraoperative visualization is performed with the SpectrumTM Fluorescence Imaging Platform (Quest Innovations, Middenmeer, The Netherlands) directly after each ICG injection assessing bowel perfusion at two different time points per anastomosis respectively: before and after anastomosis formation.

Postoperative NIRF-perfusion rate assessment Using the Quest Research SoftwareTM, the recordings before and after anastomosis formation will be analysed for their perfusion rate. This analysis will provide objective, quantitative data on the perfusion for a certain time frame which is determined by the length of the video recording. This data will be collected for statistical analysis and correlation with anastomotic leak as well as postoperative outcome.

Clinical data and follow-up Clinical data will be collected from all patients regarding anastomotic leak, bowel ischemia and necrosis as well as 30 day postoperative morbidity, mortality and length and cost of hospital stay.

Further data analysis will be performed using Microsoft Excel® and IBM SPSS®.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* capability of signing informed consent
* diagnosis of malignancies of the upper gastrointestinal tract (GI), or malignancies of the lower GI, or malignancies of the hepatobiliary system, refractory ulcerative colitis, or Crohn's disease, or acute, inflammatory, degenerative functional or anatomical disorders
* Surgery possible and medically indicated to the diagnosis (esophageal resection, or subtotal or total gastrectomy, or Y-Roux reconstruction, or right or left colonic interposition, or small bowel segment resection, or ileocecal resection, or colectomy, or proctectomy with restorative ileoanal pouch (one or two-stage), or left or right hemicolectomy, or sigmoid resection, or rectal resection (deep anterior resection (TAR)), or proctectomy with colo-anal anastomosis, or abdominoperineal resection, or stoma closure, or pancreaticoduodenectomy

Exclusion Criteria:

* liver disfunction (MELD score > 10)
* ICG (indocyanine green) specific exclusion criteria as per literature (intolerance to indocyanine green or sodium iodide, iodine allergy, hyperthyroidism, autonomous thyroid adenoma, focal or diffuse autonomies of the thyroid, previously badly tolerated injection of ICG)
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
anastomotic leak | 30 days
  number of patients suffering from an anastomotic leak within 30 days of operation

SECONDARY OUTCOMES:
Operative and post-operative complications | 30 days
  Clavien-Dindo for complication-level classification
Length of hospital stay | 100 days
  length in days

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Campus Benjamin Franklin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kassis ES, Kosinski AS, Ross P Jr, Koppes KE, Donahue JM, Daniel VC. Predictors of anastomotic leak after esophagectomy: an analysis of the society of thoracic surgeons general thoracic database. Ann Thorac Surg. 2013 Dec;96(6):1919-26. doi: 10.1016/j.athoracsur.2013.07.119. Epub 2013 Sep 24. PMID 24075499
- [Background] McDermott FD, Heeney A, Kelly ME, Steele RJ, Carlson GL, Winter DC. Systematic review of preoperative, intraoperative and postoperative risk factors for colorectal anastomotic leaks. Br J Surg. 2015 Apr;102(5):462-79. doi: 10.1002/bjs.9697. Epub 2015 Feb 19. PMID 25703524
- [Background] van den Bos J, Jongen ACHM, Melenhorst J, Breukink SO, Lenaerts K, Schols RM, Bouvy ND, Stassen LPS. Near-infrared fluorescence image-guidance in anastomotic colorectal cancer surgery and its relation to serum markers of anastomotic leakage: a clinical pilot study. Surg Endosc. 2019 Nov;33(11):3766-3774. doi: 10.1007/s00464-019-06673-6. Epub 2019 Feb 1. PMID 30710314
- [Background] van den Bos J, Al-Taher M, Schols RM, van Kuijk S, Bouvy ND, Stassen LPS. Near-Infrared Fluorescence Imaging for Real-Time Intraoperative Guidance in Anastomotic Colorectal Surgery: A Systematic Review of Literature. J Laparoendosc Adv Surg Tech A. 2018 Feb;28(2):157-167. doi: 10.1089/lap.2017.0231. Epub 2017 Nov 6. PMID 29106320
- [Background] Degett TH, Andersen HS, Gogenur I. Indocyanine green fluorescence angiography for intraoperative assessment of gastrointestinal anastomotic perfusion: a systematic review of clinical trials. Langenbecks Arch Surg. 2016 Sep;401(6):767-75. doi: 10.1007/s00423-016-1400-9. Epub 2016 Mar 11. PMID 26968863